CLINICAL TRIAL: NCT03241056
Title: Increasing Memory Confidence: a Novel Intervention for Obsessive-Compulsive Disorder
Brief Title: Cognitive Checking Intervention for Maladaptive Beliefs About Memory
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding used up; recruitment slow.
Sponsor: University of Manitoba (Other)
Responsible Party: Principal Investigator, Gillian Alcolado, Assistant Professor, University of Manitoba
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H2017:142
Record Dates: First submitted 2017-07-27; First posted 2017-08-07 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2024-06

CONDITIONS: Obsessive-Compulsive Disorder
MeSH Terms: conditions — Obsessive-Compulsive Disorder | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CBT for Maladaptive Beliefs about Memory (Experimental): Using cognitive-behavioural therapy principles, this therapy is intended to examine and change maladaptive beliefs about memory as they pertain to compulsive checking.
  Interventions: Behavioral: CBT for Maladaptive Beliefs about Memory
- Treatment as Usual (Active Comparator): This is a control treatment, Treatment as Usual (TAU), which is what patients or community members would otherwise normally receive.
  Interventions: Other: Treatment as Usual

INTERVENTIONS:
Behavioral: CBT for Maladaptive Beliefs about Memory — The novel intervention is a manualized 2-session cognitive behavioural therapy. Agenda elements, including psycho-education, discussion prompts, and homework exercises are standardized across participants. In session 1, participants are taught about the cognitive theory of checking, the research support behind this theory, and how it may apply to their own checking behavior. A homework exercise is introduced and practiced to test out this theory. In session 2, the homework results are reviewed. Further education is shared on the nature of memory and the relationship to checking, and a discussion regarding how this applies to the participant's checking then takes place. A second homework exercise is introduced to test this theory.
  Arms: CBT for Maladaptive Beliefs about Memory
Other: Treatment as Usual — Treatment as Usual (TAU) during patients' time on our waitlist in our clinic will depend on at what point they have been recruited. It may consist of a 2-session group psychoeducational intervention on anxiety, any medications prescribed by their referring physicians, and/or independent therapy/counseling they may be seeking on the side. TAU for community participants will include any treatments they are currently seeking. Information about participation in such interventions will be collected during the course of the study (at each assessment visit) in order to accurately characterize participants' TAU in the current study.
  Arms: Treatment as Usual

SUMMARY:
A small (N = 24) pilot study developed a new and brief cognitive-behavioural therapy (CBT) module for checking symptoms (CBT-C) in obsessive-compulsive disorder (OCD). CBT-C targets maladaptive beliefs about memory and results show that it is effective at significantly decreasing checking symptoms as compared to a waitlist control. The objectives of the current investigation are to further investigate CBT-C by (1) replicating the pilot results in a larger sample; (2) using an active control condition (treatment as usual) as the comparison condition (3) including a 6-month follow-up, and (4) determining whether the association between maladaptive beliefs about memory at pre-treatment assessment are related to degree of checking symptom reduction following CBT-C. The findings of the study will have theoretical significance in adding to our understanding of the maladaptive belief domains relevant to the development and maintenance of OCD and supporting the cognitive model of compulsive checking. The relevant clinical significance is the further development of an intervention that could improve outcomes in treatment of persons with OCD. The key practical outcome of the research would be to add a stepped care offering to patients with OCD.

ELIGIBILITY:
Inclusion Criteria:

* Adult over the age of 18 living in the province of Manitoba, Canada.
* Diagnosis of OCD with clinically significant levels of compulsive checking (i.e., able to meet the diagnostic criteria for OCD according to the Diagnostic and Statistical Manual of Mental Disorders, 5th Edition based solely on checking symptoms. Other OCD symptoms may be present and checking does not need to be the primary symptom.)

Exclusion Criteria:

* Active psychosis
* Active Mania
* Presence of a substance use disorder that would interfere with participation in the treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2018-01-04 (Actual); Primary Completion 2023-07-28 (Actual); Study Completion 2023-07-28 (Actual)

PRIMARY OUTCOMES:
Vancouver Obsessional Compulsive Inventory - checking subscale (change) | Change in checking symptoms from pre-treatment to post-treatment at 3 weeks later
  This six-item subscale of a self-report questionnaire measure assesses severity of checking-related OCD symptoms.
Average time spent checking per week (change) | Change in average time spent checking from pre-treatment to post-treatment at 3 weeks later
  Participants record their daily time spent checking in daily diary records while in the active phase of the study.
Vancouver Obsessional Compulsive Inventory - checking subscale | Avarege time spent checking at 6-month follow-up
  This six-item subscale of a self-report questionnaire measure assesses severity of checking-related OCD symptoms.

SECONDARY OUTCOMES:
Beliefs about Memory Inventory (change) | Change in beliefs about memory from pre-treatment to post-treatment at 3 weeks later
  Self-report questionnaire that assesses extent participant believes they have a bad memory.
Beliefs about Memory Inventory | Beliefs about memory at 6 month follow-up
  Self-report questionnaire that assesses extent participant believes they have a bad memory.
Obsessive Beliefs Questionnaire (change) | Change in obsessive beliefs from pre-treatment to post-treatment at 3 weeks later
  Self-report questionnaire that assesses maladaptive belief domains known to be related to checking. The responsibility/threat subscale is of particular interest as it is known to be related to checking behaviour.
Obsessive Beliefs Questionnaire | Obsessive beliefs at 6-month follow-up
  Self-report questionnaire that assesses maladaptive belief domains known to be related to checking. The responsibility/threat subscale is of particular interest as it is known to be related to checking behaviour.

CONTACTS AND LOCATIONS:
Locations (1):
- St. Boniface Hospital, Winnipeg, Manitoba, Canada

IPD SHARING:
Plan to Share IPD: No